CLINICAL TRIAL: NCT07147322
Title: The Effect of Basic Life Support Training in a Virtual Environment on Perceived Stress and Measured Stress Responses Compared to Conventional Basic Life Support Training
Brief Title: Virtual vs. Traditional CPR Training: Effects on Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Pasi Lehto, Medical doctor, Clinical lecturer, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 162/2024
Record Dates: First submitted 2025-08-12; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Heart Rate Variability, Biomarker of Stress; Stress and Anxiety
Keywords: heart rate variability; perceived mental workload; Virtual reality; Medical education; Basic life support
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will assigned to receive basic life support education either face to face (traditional) or in virtual reality environment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Face-to-face Basic Life Support educational training (Other): Traditional face-to-face Basic Life Support training for undergraduate medical students. Education based on European resuscitation council guidelines. Education period includes info and session lasting aprox. 30min/participant.
  Interventions: Other: Medical education, basic life support training
- Basic Life Support training for undergraduate medical students in virtual reality environment (Other): Basic Life Support training for undergraduate medical students in virtual reality environment. Education based on European resuscitation council guidelines. Education period includes info and session lasting aprox. 30min/participant.
  Interventions: Other: Medical education, basic life support training

INTERVENTIONS:
Other: Medical education, basic life support training — One basic life support training session / participant. Duration of educational session aprox. 30min.
  Other Names: face to face basic life support training; basic life support training in virtual reality environment

SUMMARY:
This medical education study investigates stress levels among undergraduate medical students during basic life support (BLS) training. It compares traditional face-to-face teaching session with virtual reality (VR) training simulating a resuscitation scenario in a public place. We will measure heart rate, heart rate variability, and self-reported stress to assess acute stress responses. The study also examines physical sensations related to VR, the realism of the virtual environment, and the suitability of VR for BLS training.

DETAILED DESCRIPTION:
Cardiac arrest is a major cause of mortality, with survival depending heavily on timely and effective cardiopulmonary resuscitation (CPR). Basic life support (BLS) training teaches recognition of cardiac arrest, calling for help, providing chest compressions and ventilations, and using an automated external defibrillator (AED). For healthcare students, regular BLS training is essential but often limited by time, resources, and staff availability. Simulation-based training provides safe practice opportunities, but traditional methods can be resource-intensive.

Virtual reality (VR) offers an alternative, enabling immersive, interactive training with lower resource requirements. VR can simulate realistic resuscitation scenarios in varied environments, potentially increasing engagement, situational awareness, and learning outcomes. However, VR may also induce physical symptoms such as nausea or dizziness, and its effectiveness compared with conventional training remains under investigation.

This pilot study compares conventional face-to-face BLS training with VR-based training delivered via head-mounted displays simulating a public cardiac arrest. The primary objective is to evaluate stress responses between the two methods, measured physiologically by heart rate variability (HRV) and psychologically by validated stress and workload questionnaires. Secondary objectives are to assess VR-related physical symptoms, the perceived realism and usability of the VR environment, and its suitability as a BLS teaching method.

The VR environment replicates a public setting with bystanders and distractions. Compressions are performed on a manikin mapped to a virtual patient, with real-time feedback on depth and rate. A virtual AED is integrated into the simulation.

Sixty first- or second-year medical students will be randomized to VR-based or conventional manikin-based BLS training (30 per group). Exclusion criteria include pregnancy, prior healthcare experience, and BLS training within the past six months. Previous VR experience will be recorded.

Physiological stress will be recorded using a three-lead surface ECG (Bittium Faros 180, Finland), providing continuous heart rate and HRV data. Approximately three hours of data will be collected, including baseline rest, training, and post-session recovery.

Participants will complete pre- and post-session questionnaires (STAI (state anxiety; NASA-TLX (task load); System Usability Scale (SUS); Simulation Sickness Questionnaire (SSQ); Simulation Design Scale (SDS): Credibility/Presence measures) All surveys will be completed electronically. A standard debrief follows each session.

The study is approved by the regional ethics committee and conducted under GDPR and the Declaration of Helsinki. Participation is voluntary with informed consent. VR may cause mild symptoms such as nausea or dizziness; sessions will be stopped if symptoms become limiting. Data are pseudonymized and securely stored.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers (18-30 years old) will be recruited from first- and second-year medical students
* Participants must be healthy young individuals with no known heart disease, normal physical performance capacity, and no current physical limitations that would affect the ability to perform chest compressions.

Exclusion Criteria:

* Pregnant individuals will not be included
* Individuals with previous healthcare experience will not be included.
* Participants must not have received basic life support training within the past six months.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Stress and Workload Compared Between Two Basic Life Support Training Environments | During training session (approximately 2 hours, including pre/post questionnaires)
  To determine whether basic life support training in a virtual environment causes more stress and workload than conventional training. Stress will be measured using heart rate variability (HRV), and perceived mental workload will be assessed with validated questionnaires (STAI, NASA-TLX).
Stress (State-Trait Anxiety Inventory, STAI) questionary | Immediately after training
  Description: Stress levels assessed using the State-Trait Anxiety Inventory (STAI).
  Range: 20-80.
  Interpretation: Higher scores indicate greater situational anxiety/stress.
Physiological Stress (Heart Rate Variability, HRV) | During training session (approximately 2 hours/participant)
  Physiological Stress (Heart Rate Variability, HRV). Continuous three-lead ECG recording using skin-surface electrodes with the Bittium Faros 180 device.
  Parameters: Standard HRV indices (time-domain: SDNN, RMSSD; frequency domain: LF, HF, LF/HF ratio).
  Interpretation: Lower HRV (e.g. higher LF/HF ratio) indicates greater physiological stress.
Perceived Workload (NASA Task Load Index) | Immediately after training
  Questionnaire assessing workload across six dimensions (mental, physical, temporal demand, performance, effort, frustration).
  Range: 0-100.
  Interpretation: Higher scores indicate greater perceived workload.

SECONDARY OUTCOMES:
Evaluation of physical symptoms caused by virtual environment - Simulation Sickness (Simulation Sickness Questionnaire, SSQ) | Immediately after training
  The SSQ is a validated tool to assess simulator-related adverse effects (e.g., nausea, oculomotor strain, disorientation).
  Scoring: Items rated and combined into subscales (Nausea, Oculomotor, Disorientation) and a total score.
  Range: Scores scaled; higher scores indicate greater severity of simulation sickness.
  Interpretation: Higher total and subscale scores indicate stronger symptoms of simulator sickness.
Suitability of virtual environment for Basic life support training - System Usability (System Usability Scale, SUS) | Immediately after training
  To explore the suitability of a virtual learning environment for resuscitation training. 10-item questionnaire on usability, scored on a 5-point Likert scale and converted to a 0-100 scale.
  Range: 0-100.
  Interpretation: Higher scores indicate better usability
Simulation Design Quality (Simulation Design Scale, SDS) | Immediately after training
  20-item questionnaire evaluating simulation design (objectives, support, problem-solving, feedback, fidelity), rated 1-5.
  Range: 20-100 total.
  Interpretation: Higher scores indicate stronger agreement that the simulation was well designed.
Sense of Presence (Slater-Usoh-Steed Questionnaire) | Immediately after training
  Questionnaire measuring the feeling of "being there" in a virtual reality environment.
  Range: 1-7 per item; mean score calculated.
  Interpretation: Higher scores indicate a stronger sense of presence in VR.

CONTACTS AND LOCATIONS:
Overall Officials: Pasi M Lehto, Principal Investigator — Research group of Anaesthesiology, Medical Research Unit of Translational Medicine, University of Oulu, Oulu, Finland
Locations (1):
- Knoppi - Clinical Skills Centre, Faculty of Medicine, University of Oulu, Oulu, North Ostrobothnia, Finland

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside the research group because of Privacy and confidentiality concerns. Ethical approval limit the sharing of the data. Also, data protection laws in this case restrict handling and transferring identifiable health data. Moreover, participants are informed that their data will not be shared with outside researchers.

REFERENCES:
- [Background] Arthur, T., Loveland-Perkins, T., Williams, C. et al. Examining the validity and fidelity of a virtual reality simulator for basic life support training. BMC Digit Health 2023. https://doi.org/10.1186/s44247-023-00016-1
- [Background] Barbadoro P, Brunzini A, Dolcini J, Formenti L, Luciani A, Messi D, Papetti A, Ponzio E, Germani M; Starlab Working Collaborative Group; Adrario E. Stress responses in high-fidelity simulation and standard simulation training among medical students. BMC Med Educ. 2023 Feb 17;23(1):116. doi: 10.1186/s12909-023-04101-x. PMID 36797725